CLINICAL TRIAL: NCT06226272
Title: Clinical Outcome Measure at Stryker Spine: COMPASS
Brief Title: Clinical Outcome Measure at Stryker Spine
Acronym: COMPASS
Status: Not yet recruiting | Type: Observational
Sponsor: Stryker Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: S-S-102
Record Dates: First submitted 2024-01-04; First posted 2024-01-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Degenerative Disc Disease; Degenerative Scoliosis
Keywords: Device: Cervical or Thoracolumbar Spinal fusion; Device: Adult Spinal Deformities
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- S-S-102-A: Cervical Sub-Protocol: The study population includes subjects who are surgically treated with a Stryker device for a cervical condition per the specific device cleared IFUs and Surgical Technique Guides (STGs), by a participating investigator and are willing to complete patient-reported questionnaires at the study-specific time points.
  Interventions: Device: Spinal Fusion
- S-S-102-B: Thoracolumbar Sub-Protocol: The study population includes subjects who are surgically treated with a Stryker device for a thoracic/lumbar condition per the specific device cleared IFUs and STGs, by a participating investigator and are willing to complete patient-reported questionnaires at the study-specific time points.
  Interventions: Device: Spinal Fusion
- S-S-102-C: Adult Spinal Deformities: The study population includes subjects who are surgically treated with a Stryker device for a spinal deformity condition per the specific device cleared IFUs and STGs, by a participating investigator and are willing to complete patient-reported questionnaires at the study-specific time points.
  Interventions: Device: Spinal Deformities Correction

INTERVENTIONS:
Device: Spinal Fusion — Cervical Spinal Fusion
  Groups: S-S-102-A: Cervical Sub-Protocol
Device: Spinal Fusion — Thoracic / Lumbar Spinal Fusion
  Groups: S-S-102-B: Thoracolumbar Sub-Protocol
Device: Spinal Deformities Correction — Spinal Deformities Correction
  Groups: S-S-102-C: Adult Spinal Deformities

SUMMARY:
This is a multicenter, prospective, retrospective, Post Market Clinical Follow-up (PMCF) study in subjects who have undergone or will undergo surgery utilizing one or more Stryker devices according to Stryker cleared Instructions for Use (IFU).

DETAILED DESCRIPTION:
Stryker Spine has a broad portfolio of spinal devices used to stabilize the spine. This PMCF study is designed to collect data on the performance and safety of the devices over their lifetime of 24 months post-implantation. Four protocols have been designed to aid in this process, a master and three sub-protocols. The sub-protocols are based on body region and indication:

* S-S-102-A Cervical: Interbody Devices (IBDs), Vertebral Body Replacement Devices (VBRs), Internal Fixation Devices, and Vitoss
* S-S-102-B Thoracolumbar: IBDs, VBRs, Internal Fixation Devices, and Vitoss
* S-S-102-C Adult Spinal Deformities: IBDs, Internal Fixation Devices, and Vitoss Each of the sub-protocols has its own specific performance endpoint and hypothesis, radiographical data assessments, and SAPs. Safety data will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

• To be eligible to participate in the study, the potential subject must meet all inclusion criteria specific to the Stryker system being evaluated, please contact one of the participating investigators or see the device-specific cleared IFU, for further details.

Exclusion Criteria:

• The exclusion criteria are based on the contraindications as presented in the Stryker device cleared IFUs, please contact one of the participating investigators or see the device-specific cleared IFU, for further details.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects who have undergone or will undergo surgery utilizing one or more Stryker devices according to Stryker cleared IFUs and Surgical Technique Guides (STGs) by a participating investigator and are willing to complete the following patient-reported outcome measures (PROMs) at the study-specific time points.
Sampling Method: Non-Probability Sample
Enrollment: 5222 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2029-01-29 (Estimated); Study Completion 2032-01-29 (Estimated)

PRIMARY OUTCOMES:
S-S-102-A | Baseline through 24-months post-op.
  Mean change in the subject's Neck Disability Index (NDI) score.
S-S-102-B | Baseline through 24-months post-op.
  Mean change in the subject's Oswestry Disability Index (ODI) score.
S-S-102-C | Baseline through 24-months post-op.
  Mean change in the subject's Scoliosis Research Society-22 revised (SRS-22r).

SECONDARY OUTCOMES:
S-S-102-A | Surgery through 24-months post-op.
  The incidence of the following safety events:
  * Serious Adverse Events (AEs)
  * Device-related AEs
  * Procedure-related AEs
  * Operative AEs
  * Secondary spine surgeries
S-S-102-B | Surgery through 24-months post-op.
  The incidence of the following safety events:
  * Serious Adverse Events (AEs)
  * Device-related AEs
  * Procedure-related AEs
  * Operative AEs
  * Secondary spine surgeries
S-S-102-C | Surgery through 24-months post-op.
  The incidence of the following safety events:
  * Serious Adverse Events (AEs)
  * Device-related AEs
  * Procedure-related AEs
  * Operative AEs
  * Secondary spine surgeries

IPD SHARING:
Plan to Share IPD: No